CLINICAL TRIAL: NCT05290493
Title: A Randomized, Placebo-Controlled Crossover Trial to Assess the Safety and Efficacy of NB-001 in Children and Adolescents With 22q11 Deletion Syndrome
Brief Title: NB-001 in Children and Adolescents With 22q11 Deletion Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nobias Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NB-001-01
Record Dates: First submitted 2022-01-26; First posted 2022-03-22 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: 22q11 Deletion Syndrome
Keywords: 22q11 Deletion Syndrome; 22q11.2 Deletion Syndrome; 22q11DS; Children and Adolescents
MeSH Terms: conditions — 22q11 Deletion Syndrome; DiGeorge Syndrome | interventions — 5-((2-(6-Amino-9H-purin-9-yl) ethyl) amino)-1-pentanol

STUDY DESIGN:
Intervention Model Description: Subjects were randomized in a 1:1 ratio to one of two treatment sequences: NB-001 (active drug product) followed by placebo (treatment sequence A/P) or placebo followed by NB-001 (treatment sequence P/A). Subjects received IP corresponding with their first treatment assignment for 6 weeks (Treatment Period 1), followed by an intervening wash-out period of 1 week, and then received their second treatment assignment for the subsequent 6-week period (Treatment Period 2).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: NB-001 and matching placebo were supplied to the Investigator or designee in blinded plastic bottles, each containing 40 capsules. Additionally, subject and parent/guardian, the Investigator, clinical trial site personnel, home health nurses, centralized rater(s), and the Sponsor will be blinded to treatment sequence assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NB-001 (Experimental): Two (2) 100 mg capsules administered orally BID (400 mg total daily dose) with liquids or, if the subject is unable to swallow a capsule whole, capsules were opened, and the contents sprinkled on applesauce.
  Interventions: Drug: NB-001
- Placebo (Placebo Comparator): Two (2) capsules (matching, inactive) administered orally BID with liquids or, if the subject is unable to swallow a capsule whole, capsules were opened, and the contents sprinkled on applesauce.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: NB-001 — Non-stimulant modulator of metabotropic glutamate receptors (mGluRs)
  Other Names: fasoracetam monohydrate; (5R)-5-(piperidine-1-carbonyl)pyrrolidin-2-one monohydrate
  Arms: NB-001
Other: Placebo — Matching, inactive placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, placebo-controlled crossover trial to assess the safety and efficacy of NB-001 in children and adolescents with 22q11DS that manifest commonly associated neuropsychiatric symptoms.

DETAILED DESCRIPTION:
The trial is designed to allow all visits to be conducted via telephone and/or video (i.e., telemedicine) or by home health nurse. An in-person visit is required at Screening unless site or government mandates restrict this due to coronavirus disease-2019 (COVID-19). Other in-person visit(s) may occur, if indicated, based on the Investigator's clinical judgement. Subjects will be screened to confirm eligibility and then randomized in a 1:1 ratio to one of two treatment sequences: NB-001 (active drug product) followed by placebo (treatment sequence A/P) or placebo followed by NB-001 (treatment sequence P/A). During the Double-Blind Treatment Phase of the trial, the subject and/or parent/legal guardian (henceforth, 'parent/guardian') will be contacted at Day 0 to complete baseline symptom scales and will begin dosing with the investigational product (IP; NB-001 or placebo) on the morning of Day 1. Subjects or their parent/guardian will administer the IP twice daily (BID) and will be contacted at Days 0, 1, 14, 28, 42, 49, 50, 63, 77 and 91 to evaluate measures of safety and efficacy, including the completion of symptom scales. In addition, the subject and/or parent/guardian will be contacted at Days 7, 21, 35, 56, 70 and 84 to assess subject safety. Blood samples for pharmacokinetic analysis, 4β-hydroxycholesterol and plasma proline will be collected at multiple timepoints. During the Double-Blind Treatment Phase, subjects will receive IP corresponding with their first treatment assignment for 6 weeks (Treatment Period 1), followed by an intervening wash-out period of 1 week, and then will receive their second treatment assignment for the subsequent 6-week period (Treatment Period 2). All symptom scales will be centrally and/or locally administered. Approximately 10 parents/guardians and paired clinical trial site clinicians for subjects who complete the trial per protocol through Visit Day 91 will be invited to participate in an optional, one-hour (approximately), exit interview to discuss the observations of the subject's experience(s) and functioning while participating in the treatment periods of the trial. The subject and/or parent/guardian will be contacted for an End of Trial Visit to occur 4 weeks following the last dose of IP to assess safety.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has a genotype with a pathologic deletion in the 22q11 region confirmed by documentation (e.g., genetic test results) available at the clinical trial site.
2. The subject is aged 6 to 17 years old, inclusive.
3. The subject has a CGI-S scale score of ≥4 (i.e., moderately, markedly, severely, or among the most extremely ill patients) at Screening. Note that the Severity score of 4 could be from a composite of 2 or more sub-threshold scores.

   And either:
   1. Psychiatric symptoms in the clinical range for at least 1 of 3 disorders, anxiety disorder, ADHD, or ASD, respectively, as demonstrated by score(s) at or above the following numbers on at least 1 of 3 scales:

      * PARS 5-Item Severity Score ≥12 (i.e., sum of items 2+3+5+6+7 ≥12)
      * ADHD-RS-5 Scores of 2 or 3 (i.e., "Often" or "Very Often") on at least 6 questions, with the majority of symptoms related to inattention (common in 22q11DS) rather than hyperactivity (less common in 22q11DS)
      * SRS-2 >60

      OR:
   2. Psychiatric symptoms in the subclinical range for at least 2 of 3 disorders, anxiety disorder, ADHD, and/or ASD, respectively, as demonstrated by scores at or above the following numbers on at least 2 of 3 scales:

      * PARS 5-Item Severity Score of 10 or 11 (i.e., sum of items 2+3+5+6+7=10 or 11)
      * ADHD-RS-5 Scores of 2 or 3 (i.e., "Often" or "Very Often") on 4 or 5 questions, with the majority of symptoms related to inattention (common in 22q11DS) rather than hyperactivity (less common in 22q11DS)
      * SRS-2 of 55-59
4. The subject has adequate renal and hepatic function indicated by:

   * Estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73 m2 (per the revised Schwartz equation; Fadrowski and Furth 2011, Staples et al. 2010)
   * Serum bilirubin ≤2.5 × upper limit of normal (ULN; unless documented Gilbert's Disease); aspartate aminotransferase and alanine aminotransferase ≤2.5 × ULN
5. If the subject is female and of reproductive potential, she has a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day 0.
6. If the subject is of reproductive potential, s/he agrees to abstain from reproductive cell donation, per below, and, if ever heterosexually active, to use dual effective/highly effective contraception (including at least one effective and at least one highly effective contraceptive method; Section 9.2.1) from Screening through the End of Trial Visit.

   * If the subject is female and of reproductive potential, she agrees to abstain from oocyte donation from Screening through the End of Trial Visit.
   * If the subject is male and of reproductive potential, he agrees to abstain from sperm donation from Screening through the End of Trial Visit.
7. The subject's parent/guardian understands the trial procedures and agrees to the subject's participation in the trial, as well as to the parent/guardian trial involvement, as indicated by parent/guardian signature on the informed consent form and, if applicable, subject signature on the subject assent form.

Exclusion Criteria:

1. The subject or parent/guardian is, in the opinion of the Investigator, mentally or legally incapacitated, or has significant emotional problems at the time of Screening or expected emotional problems during the conduct of the trial which would interfere with the conduct of the trial evaluations.
2. The subject has a history of psychotic symptoms, current psychotic symptoms, or a diagnosis of a psychotic disorder based on clinical assessment.
3. The subject has an intelligence quotient (IQ) score of <65 based on the WASI-II assessment. NOTE: A maximum of 3 (i.e., 10% of the total N) nonverbal subjects will be allowed in the trial on a first-come-first-served basis.
4. The subject has a history of any illness that, in the opinion of the Investigator, might confound the results of the trial or pose an additional risk to the subject by participation in the trial.
5. The subject has clinically significant unstable or uncontrolled endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases.
6. The subject has uncontrolled, active seizure(s), within the 3 months prior to Screening.
7. The subject has known human immunodeficiency virus (HIV), a detectable viral load for hepatitis C, or hepatitis B surface antigen indicative of chronic active infection.
8. The subject is pregnant or is a nursing mother.
9. The subject has suicidal ideation and behavior, based on Investigator assessment of the completed Columbia-Suicide Severity Rating Scale at Screening, or when repeated on Day 0 (if more than 21 days elapse between Screening and Day 1).
10. The subject is currently taking neuropsychiatric medication(s) at a dose that has not been stable for ≥3 months prior to Day 1 or psychotherapy that has not been stable for ≥3 months prior to Day 1. If the subject is taking medication(s) or receiving psychotherapy, the subject and parent/guardian must agree to continue the intervention(s) at the same dose and frequency through the End of Trial Visit.
11. The subject has received any investigational therapy (i.e., used for a non-approved indication and in the context of a research investigation) <14 days prior to the first dose of NB-001 (i.e., Day 1) or within 5 drug half-lives prior to the first dose of NB-001.
12. The subject uses illicit drugs (e.g., marijuana, amphetamines or cocaine), or has known alcohol or drug abuse or dependence, as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (American Psychiatric Association 2013). Medically approved marijuana use, where usage is legal, is allowed; however, the dose and frequency of use should remain stable during trial participation.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - Seattle Children's Hospital, Seattle, Washington
- The Hospital for Sick Children (SickKids), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (6 Weeks) Then Washout (1 Week) Then NB-001 (6 Weeks): Subjects received Placebo for 6 weeks (Treatment Period 1), followed by an intervening wash-out period of 1 week. Subjects then received NB-001 for the subsequent 6-week period (Treatment Period 2).
- NB-001 (6 Weeks) Then Washout (1 Week) Then Placebo (6 Weeks): Subjects received NB-001 for 6 weeks (Treatment Period 1), followed by an intervening wash-out period of 1 week. Subjects then received Placebo for the subsequent 6-week period (Treatment Period 2).
Period: Overall Study
Arm/Group | Placebo (6 Weeks) Then Washout (1 Week) Then NB-001 (6 Weeks) | NB-001 (6 Weeks) Then Washout (1 Week) Then Placebo (6 Weeks)
Started | 18 | 19
Completed | 15 | 17
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) includes all subjects who received at least one capsule of investigational product (IP). The numbers are different than the numbers of participants in the Participant Flow as the SAS excludes subjects who withdrew their participation prior to taking their first dose of IP. Thus, 1 subject in the Placebo/NB-001 group, and 2 subjects in the NB-001/Placebo group, were excluded from the SAS since they discontinued trial participation prior to taking any dose of IP.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (6 Weeks) Then Washout (1 Week) Then NB-001 (6 Weeks) | NB-001 (6 Weeks) Then Washout (1 Week) Then Placebo (6 Weeks) | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.1 (3.12) | 11.9 (3.30) | 12.0 (3.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 11 | 11 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 13 | 15 | 28
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 3 | 6
  United States | 14 | 14 | 28
Reproductive Potential [Count of Participants; unit: Participants]
  Yes | 8 | 9 | 17
  No | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of NB-001
Description: Type, frequency, severity, and causality of treatment-emergent adverse events (TEAEs),treatment-emergent serious adverse events (TESAEs), clinically significant changes from baseline in laboratory tests, electrocardiograms (ECGs), vital signs, and physical examination findings during treatment with NB-001.
Time Frame: 6 weeks (Day 42/ET)
Population: Safety Analysis Set: Includes all subjects who receive at least one capsule (100 mg) of IP.
Measure: Count of Participants; unit: Participants
Groups:
- NB-001: Active drug product, NB-001: Two (2) 100 mg capsules will be administered orally BID with liquids or, if the subject is unable to swallow a capsule whole, capsules may be opened, and the contents sprinkled on applesauce; total daily dose: 400 mg.
- Placebo: Placebo: Two (2) capsules (inactive, matching NB-001) will be administered orally BID with liquids or, if the subject is unable to swallow a capsule whole, capsules may be opened, and the contents sprinkled on applesauce.
Arm/Group | NB-001 | Placebo
Number analyzed (Participants) | 33 | 34
Participants
  Subjects Reporting at Least One TEAE | 18 | 24
  CTCAE Grade 1: Mild | 14 | 20
  CTCAE Grade 2: Moderate | 4 | 4
  CTCAE Grade 3: Severe | 0 | 0
  CTCAE Grade 4: Life-threatening | 0 | 0
  CTCAE Grade 5: Causing Death | 0 | 0
  TEAE Relationship: Not Related | 12 | 20
  TEAE Relationship: Related | 6 | 4
  TEAE Leading to Discontinuation of IP | 0 | 1
  TEAE Requiring Temporary Dose Interruption of IP | 1 | 0
  TEAE Requiring Dose Reduction of IP | 0 | 1
  TEAE Leading to Premature Withdrawal from the Study | 0 | 1
  TEAE of Special Interest | 2 | 0
  TEAE Causing Death | 0 | 0
  Subjects Reporting at Least One TESAE | 0 | 0

2. Secondary Outcome: Treatment Effect of NB-001 on the Clinical Global Impression Improvement (CGI-I) Scale
Description: The CGI-I scale is a 7-point scale that measures how much a patient's condition has improved or worsened over time. The CGI-I is scored on a scale of 1-7, with a score of 1 indicating "Very much improved" and 7 indicating "Very much worse". The least squares mean of the score on the CGI-I scale at the end of the 6-week treatment period is reported here.
Time Frame: 6 weeks (Day 42/ET)
Population: Full Analysis Set (FAS): Includes all subjects in the Enrolled Analysis Set (those who meet all eligibility criteria and consent to participate in study) who have at least one valid post-baseline efficacy evaluation within each treatment period. Subjects are analyzed based on the treatment to which they were randomized in each treatment period.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | NB-001 | Placebo
Number analyzed (Participants) | 33 | 33
Score on a scale | 3.34 (0.154) | 3.69 (0.154)
Statistical Analysis 1: Comparison: NB-001 vs Placebo; Test type: Superiority; p = 0.0672, Mixed Models Analysis

3. Secondary Outcome: Treatment Effect of NB-001 on the Clinical Global Impression Severity (CGI-S) Scale
Description: CGI-S: 7-point scale that measures a participant's overall disease severity. A 1-point improvement in the CGI-S scale is an appropriate meaningful change threshold. Possible scores are: 1 = Normal, not at all impaired; 2 = Borderline impaired; 3 = Mildly impaired; 4 = Moderately impaired; 5 = Markedly impaired; 6 = Severely impaired; 7 = Among the most extremely impaired patients.
Time Frame: 6 weeks (Day 42/ET)
Population: Full Analysis Set: Includes all subjects in the Enrolled Analysis Set (those who meet all eligibility criteria and consent to participate in study) who have at least one valid post-baseline efficacy evaluation within each treatment period. Subjects are analyzed based on the treatment to which they were randomized in each treatment period.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | NB-001 | Placebo
Number analyzed (Participants) | 33 | 33
score on a scale | 4.14 (0.121) | 4.12 (0.121)
Statistical Analysis 1: Comparison: NB-001 vs Placebo; Test type: Superiority; p = 0.2045, Mixed Models Analysis

4. Secondary Outcome: Treatment Effect of NB-001 on the Pediatric Anxiety Rating Scale (PARS)
Description: The PARS is a clinician-rated instrument for assessing severity of anxiety symptoms associated with common anxiety disorders. The first section is a 50-item symptom checklist and the second section is comprised of 7 severity/impairment items reflecting the severity/impairment of all symptoms noted in the first section.
  The PARS total severity score is calculated as the sum of items 2, 3, 5, 6, and 7 from the second section of the instrument. Each item is rated on a 6-point Likert scale from 0-5 with the higher scores indicating more severe anxiety. The total severity score can range from a minimum value of 0 to a maximum value of 25. Higher scores indicate more severe anxiety.
  Additionally, per protocol, at baseline, a score of >12 on the PARS 5-item total severity score (items 2+3+5+6+7) is indicative of psychiatric symptoms in the clinical range for anxiety disorder, and a score of 10 or 11 is indicative of psychiatric symptoms in the subclinical range for anxiety disorder.
Time Frame: 6 weeks (Day 42/ET)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | NB-001 | Placebo
Number analyzed (Participants) | 33 | 33
score on a scale | 7.18 (0.728) | 8.14 (0.729)
Statistical Analysis 1: Comparison: NB-001 vs Placebo; Test type: Superiority; p = 0.2931, Mixed Models Analysis

5. Secondary Outcome: Treatment Effect of NB-001 on the Attention Deficit Hyperactivity Disorder-Rating Scale (ADHD-RS-5) - Inattention Score
Description: The ADHD-RS-5 is a parent/guardian reported scale to measure behaviors of children and adolescents with ADHD. It consists of 18 items grouped into two subscales: inattention (items 1-9) and hyperactivity (items 10-18). Each item is scored on a scale ranging from 0 (reflecting no symptoms) to 3 (reflecting severe symptoms). The total inattention score (reported here) can range from a minimum value of 0 to a maximum value of 27. Higher total inattention scores reflect more severe symptoms.
Time Frame: 6 weeks (Day 42/ET)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | NB-001 | Placebo
Number analyzed (Participants) | 33 | 33
score on a scale | 13.47 (0.947) | 13.80 (0.941)
Statistical Analysis 1: Comparison: NB-001 vs Placebo; Test type: Superiority; p = 0.7799, Mixed Models Analysis

6. Secondary Outcome: Treatment Effect of NB-001 on the Attention Deficit Hyperactivity Disorder-Rating Scale (ADHD-RS-5) - Hyperactivity Score
Description: The ADHD-RS-5 is a parent/guardian reported scale to measure behaviors of children and adolescents with ADHD. It consists of 18 items grouped into two subscales: inattention (items 1-9) and hyperactivity (items 10-18). Each item is scored on a scale ranging from 0 (reflecting no symptoms) to 3 (reflecting severe symptoms). The total hyperactivity score (reported here) can range from a minimum value of 0 to a maximum value of 27. Higher total hyperactivity scores reflect more severe symptoms.
Time Frame: 6 weeks (Day 42/ET)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | NB-001 | Placebo
Number analyzed (Participants) | 33 | 33
score on a scale | 7.82 (0.629) | 8.02 (0.623)
Statistical Analysis 1: Comparison: NB-001 vs Placebo; Test type: Superiority; p = 0.7974, Mixed Models Analysis

7. Secondary Outcome: Treatment Effect of NB-001 on the Social Responsiveness Scale, Second Edition (SRS-2)
Description: The SRS-2 identifies the presence and severity of social impairment within the autism spectrum. It is a 65-item, parent-completed questionnaire which incorporates 5 content areas of social deficits. The sum of all items is calculated to provide a maximum total score of 195. However, a total derived T-score is calculated centrally and reported for this trial. A higher T-score indicates more severe impairment. The population mean T-score is 50, with a standard deviation of 10. Thus, a T-score considered within the normal range is 59 or below (i.e., minimum T-score value), and a T-score indicating a severe range is 76 or above (i.e., maximum T-score value). Scores between 60-75 fall into the mild to moderate range.
Time Frame: 6 weeks (Day 42/ET)
Population: Includes all subjects in the Enrolled Analysis Set (those who meet all eligibility criteria and consent to participate in study) who have at least one valid post-baseline efficacy evaluation within each treatment period. Subjects are analyzed based on the treatment to which they were randomized in each treatment period.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | NB-001 | Placebo
Number analyzed (Participants) | 33 | 33
T-score | 62.42 (1.005) | 63.27 (1.019)
Statistical Analysis 1: Comparison: NB-001 vs Placebo; Test type: Superiority; p = 0.8286, Mixed Models Analysis

8. Other Pre Specified Outcome: Exit Interview
Description: Optional qualitative exit interviews were conducted with clinicians and parent/guardian(s) of subjects who completed the protocol.
Time Frame: End of Treatment; approximately 13 weeks of trial participation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Approximately 21 weeks: Adverse Events (AEs) were collected from the time of signing the Informed Consent Form (ICF) to the End of Trial Visit (Day 119).
Description: Treatment-emergent AEs are defined as those AEs with onset after the first dose of IP or existing events that worsened after the first dose during the study. Any AE that occurred between the date of ICF signature and the date/time of first IP administration was considered a pre-treatment-emergent AE. At each level of summarization (any event, system organ class, and preferred term), subjects reporting more than one AE are counted only once.
Groups:
- NB-001: Active drug product, NB-001: Two (2) 100 mg capsules administered orally BID with liquids or, if the subject is unable to swallow a capsule whole, capsules may be opened, and the contents sprinkled on applesauce; total daily dose: 400 mg.
  NB-001: NB-001 is a non-stimulant modulator of multiple metabotropic glutamate receptors (mGluRs).
- Placebo: Placebo: Two (2) capsules (matching NB-001) administered orally BID with liquids or, if the subject is unable to swallow a capsule whole, capsules may be opened, and the contents sprinkled on applesauce.
  Placebo: Matching, inactive placebo
Arm/Group | NB-001 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 18/33 | 24/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NB-001 (N=33) | Placebo (N=34)
Nasopharyngitis (Infections and infestations) | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Insomnia (Psychiatric disorders) | 1 | 6
Irritability (Psychiatric disorders) | 1 | 3
Anxiety (Psychiatric disorders) | 1 | 2
Panic attack (Psychiatric disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Fatigue (General disorders) | 3 | 1 — General disorders and administration site conditions
Pyrexia (General disorders) | 2 | 2 — General disorders and administration site conditions
Headache (Nervous system disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/93/NCT05290493/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT05290493/SAP_001.pdf